CLINICAL TRIAL: NCT00798616
Title: Are Steroids Efficacious in Hospitalized Patients With Bronchiolitis Who Show an Objective Clinical Improvement After Albuterol ("Albuterol Responders")?
Brief Title: Steroids Helping Albuterol Responders Exclusively
Acronym: SHARE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to enroll a sufficient number of patients due to manpower.
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Steven Shein, Chief Resident, Department of Pediatrics, University Hospitals of Cleveland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHC 07-08-36
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2010-10

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; steroids; corticosteroids; albuterol; child; infant; pediatric
MeSH Terms: conditions — Bronchiolitis | interventions — Prednisolone; Methylprednisolone; Adrenal Cortex Hormones; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Responders/Placebo (Placebo Comparator): Albuterol responders being given placebo
  Interventions: Drug: placebo
- Responders/Steroids (Active Comparator): albuterol responders being given steroids
  Interventions: Drug: prednisolone or methylprednisolone
- Non-responders/placebo (Placebo Comparator): non-albuterol responders being given placebo
  Interventions: Drug: placebo
- non-responders/steroids (Active Comparator): non-albuterol responders being given steroids
  Interventions: Drug: prednisolone or methylprednisolone

INTERVENTIONS:
Drug: prednisolone or methylprednisolone — either prednisolone 2mg/kg PO once daily or methylprednisolone 1.6mg/kg IV once daily (if IV access is present) for length of hospitalization, for a maximum of seven days
  Other Names: corticosteroids; Solu-Medrol; Orapred
  Arms: Responders/Steroids; non-responders/steroids
Drug: placebo — oral or IV placebo
  Arms: Non-responders/placebo; Responders/Placebo

SUMMARY:
The purpose of the study is to determine whether corticosteroids are beneficial to children with bronchiolitis whose breathing gets better after being given a breathing treatment with albuterol.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bronchiolitis
* Respiratory Distress Assessment Index score of 4 or more

Exclusion Criteria:

* prior prescription of bronchodilators or inhaled corticosteroids
* birth at <36 weeks gestation
* chronic cardiac disease
* chronic pulmonary disease (including asthma)
* immunodeficiency
* non-topical steroid use in the prior week
* parents that don't understand English
* baseline systolic blood pressure >118 mmHg
* home oxygen use
* evidence of systemic fungal or varicella infection
* bronchodilator use in the prior week
* allergy to albuterol or corticosteroids

Ages: 4 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
respiratory rate and respiratory distress score | 4 hours
length of hospitalization (actual and until meets "ready for discharge" criteria) | variable, likely no more than 2 weeks

SECONDARY OUTCOMES:
need for increased respiratory support (intubation, CPAP, BiPAP) | variable, likely up to 2 weeks
amount of oxygen used during hospitalization | variable, likely less than 2 weeks
number of doses of bronchodilators used during hospitalization | variable, likely no more than 2 weeks
total duration of symptoms | variable, likely no more than 3 weeks
need for unanticipated medical care after discharge | variable, likely no more than 3 weeks
tachycardia and/or hypertension during hospitalization | variable, likely no more than 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Shein, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Background] American Academy of Pediatrics Subcommittee on Diagnosis and Management of Bronchiolitis. Diagnosis and management of bronchiolitis. Pediatrics. 2006 Oct;118(4):1774-93. doi: 10.1542/peds.2006-2223. PMID 17015575
- [Background] Shay DK, Holman RC, Newman RD, Liu LL, Stout JW, Anderson LJ. Bronchiolitis-associated hospitalizations among US children, 1980-1996. JAMA. 1999 Oct 20;282(15):1440-6. doi: 10.1001/jama.282.15.1440. PMID 10535434
- [Background] Stang P, Brandenburg N, Carter B. The economic burden of respiratory syncytial virus-associated bronchiolitis hospitalizations. Arch Pediatr Adolesc Med. 2001 Jan;155(1):95-6. doi: 10.1001/archpedi.155.1.95. No abstract available. PMID 11177073
- [Background] Wang EE, Law BJ, Boucher FD, Stephens D, Robinson JL, Dobson S, Langley JM, McDonald J, MacDonald NE, Mitchell I. Pediatric Investigators Collaborative Network on Infections in Canada (PICNIC) study of admission and management variation in patients hospitalized with respiratory syncytial viral lower respiratory tract infection. J Pediatr. 1996 Sep;129(3):390-5. doi: 10.1016/s0022-3476(96)70071-9. PMID 8804328
- [Background] Schweich PJ, Hurt TL, Walkley EI, Mullen N, Archibald LF. The use of nebulized albuterol in wheezing infants. Pediatr Emerg Care. 1992 Aug;8(4):184-8. doi: 10.1097/00006565-199208000-00003. PMID 1513726
- [Background] Kristjansson S, Lodrup Carlsen KC, Wennergren G, Strannegard IL, Carlsen KH. Nebulised racemic adrenaline in the treatment of acute bronchiolitis in infants and toddlers. Arch Dis Child. 1993 Dec;69(6):650-4. doi: 10.1136/adc.69.6.650. PMID 8285776
- [Background] Gadomski AM, Bhasale AL. Bronchodilators for bronchiolitis. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD001266. doi: 10.1002/14651858.CD001266.pub2. PMID 16855963
- [Background] Dobson JV, Stephens-Groff SM, McMahon SR, Stemmler MM, Brallier SL, Bay C. The use of albuterol in hospitalized infants with bronchiolitis. Pediatrics. 1998 Mar;101(3 Pt 1):361-8. doi: 10.1542/peds.101.3.361. PMID 9480998
- [Background] Patel H, Platt R, Lozano JM, Wang EE. Glucocorticoids for acute viral bronchiolitis in infants and young children. Cochrane Database Syst Rev. 2004;(3):CD004878. doi: 10.1002/14651858.CD004878. PMID 15266547
- [Background] Garrison MM, Christakis DA, Harvey E, Cummings P, Davis RL. Systemic corticosteroids in infant bronchiolitis: A meta-analysis. Pediatrics. 2000 Apr;105(4):E44. doi: 10.1542/peds.105.4.e44. PMID 10742365
- [Background] Kuzik BA, Al-Qadhi SA, Kent S, Flavin MP, Hopman W, Hotte S, Gander S. Nebulized hypertonic saline in the treatment of viral bronchiolitis in infants. J Pediatr. 2007 Sep;151(3):266-70, 270.e1. doi: 10.1016/j.jpeds.2007.04.010. Epub 2007 Jun 29. PMID 17719935
- [Background] Leader S, Kohlhase K. Recent trends in severe respiratory syncytial virus (RSV) among US infants, 1997 to 2000. J Pediatr. 2003 Nov;143(5 Suppl):S127-32. doi: 10.1067/s0022-3476(03)00510-9. PMID 14615711
- [Background] Rodriguez WJ, Gruber WC, Groothuis JR, Simoes EA, Rosas AJ, Lepow M, Kramer A, Hemming V. Respiratory syncytial virus immune globulin treatment of RSV lower respiratory tract infection in previously healthy children. Pediatrics. 1997 Dec;100(6):937-42. doi: 10.1542/peds.100.6.937. PMID 9374560
- [Background] Hartling L, Wiebe N, Russell K, Patel H, Klassen TP. A meta-analysis of randomized controlled trials evaluating the efficacy of epinephrine for the treatment of acute viral bronchiolitis. Arch Pediatr Adolesc Med. 2003 Oct;157(10):957-64. doi: 10.1001/archpedi.157.10.957. PMID 14557155
- [Background] Wainwright C, Altamirano L, Cheney M, Cheney J, Barber S, Price D, Moloney S, Kimberley A, Woolfield N, Cadzow S, Fiumara F, Wilson P, Mego S, VandeVelde D, Sanders S, O'Rourke P, Francis P. A multicenter, randomized, double-blind, controlled trial of nebulized epinephrine in infants with acute bronchiolitis. N Engl J Med. 2003 Jul 3;349(1):27-35. doi: 10.1056/NEJMoa022226. PMID 12840089
- [Background] Tal A, Levy N, Bearman JE. Methylprednisolone therapy for acute asthma in infants and toddlers: a controlled clinical trial. Pediatrics. 1990 Sep;86(3):350-6. PMID 2201941
- [Background] Connett GJ, Warde C, Wooler E, Lenney W. Prednisolone and salbutamol in the hospital treatment of acute asthma. Arch Dis Child. 1994 Mar;70(3):170-3. doi: 10.1136/adc.70.3.170. PMID 8135557
- [Background] Smith M, Iqbal S, Elliott TM, Everard M, Rowe BH. Corticosteroids for hospitalised children with acute asthma. Cochrane Database Syst Rev. 2003;2003(2):CD002886. doi: 10.1002/14651858.CD002886. PMID 12804441
- [Background] Gorelick MH, Shaw KN, Murphy KO. Validity and reliability of clinical signs in the diagnosis of dehydration in children. Pediatrics. 1997 May;99(5):E6. doi: 10.1542/peds.99.5.e6. PMID 9113963